CLINICAL TRIAL: NCT02577991
Title: A Prospective, Randomized Controlled Trial on the Effect of Local Steroid Application on a Cervical Plate Versus Intravenous Steroids on Dysphagia Following Anterior Cervical Discectomy and Fusion (ACDF)
Brief Title: Effect of Local Steroid Application on a Cervical Plate Versus Intravenous Steroids on Dysphagia Following Anterior Cervical Discectomy and Fusion (ACDF)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Alpesh A. Patel, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU00085674
Record Dates: First submitted 2015-10-12; First posted 2015-10-16 (Estimated); Results first posted 2019-05-30 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Cervical Spine
MeSH Terms: interventions — Calcium Dobesilate; Triamcinolone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control group (No Intervention): No steroid
- IV steroid (Experimental): 10 mg of intraoperative intravenous decadron with gel foam sponge placed on cervical plate
  Interventions: Drug: Decadron
- Local steroid (Experimental): 40 mg of triamcinolone on gel foam sponge dabbed on the anterior cervical plate
  Interventions: Drug: Triamcinolone

INTERVENTIONS:
Drug: Decadron — 10 mg of intraoperative intravenous decadron with gel foam sponge placed on cervical plate
  Arms: IV steroid
Drug: Triamcinolone — 40 mg of triamcinolone on gel foam sponge dabbed on the anterior cervical plate
  Arms: Local steroid

SUMMARY:
Local application of steroids in ACDF surgery will lead to decreased incidence of dysphagia compared to intravenous steroids or a control group

DETAILED DESCRIPTION:
Dysphagia is a common complication after ACDF. PSTS is also a natural sequela of ACDF and can lead to airway compromise among other complications. Previous studies have demonstrated that administration of intravenous methylprednisolone (1mg/kg) after anterior cervical spine surgery reduced the incidence of pharyngolaryngeal lesions as identified by nasofibroscopic examination. Lee et al. prospectively evaluated 50 patients and determined that local application of steroids in the retropharyngeal area following ACDF reduced PSTS and odynophagia as measured by the Visual Analogue Scale (VAS) and the Neck Disability Index (NDI) compared to a control group. Furthermore, there were no adverse events/reactions from local application of steroid on a gel foam sponge in the setting of anterior spinal surgery. There are no studies in the current literature that investigate the incidence of dysphagia with application of local steroids after ACDF, nor are there any studies that stratify the efficacy of local steroids compared to intravenous steroids. There is also no current spine literature that directly compares the efficacy of intravenous steroids versus local steroids in the incidence of dysphagia or dysphonia. Our study will be the first in the literature to assess the efficacy of local steroids in reducing the incidence of dysphagia after anterior cervical spine surgery, and as a result, may improve patient outcomes after ACDF.

Dysphagia and dysphonia are common complications after anterior cervical spine surgery. Despite their clinical importance, studies on the treatment and/or prevention of these complications are limited due to the lack of valid and reliable outcome measures. The majority of research is found in the otolaryngology literature and has focused on disease pathophysiology, diagnosis, and therapy.

The Bazaz score has been used in the spine literature to evaluate dysphagia after anterior cervical discectomy and fusion (ACDF). This is a subjective questionnaire that has not been validated in the literature. Additionally, new patient-centered outcome measures, the Eating Assessment Tool (EAT-10) and Voice Handicap Index (VHI-10) have recently been developed, and in addition to the Bazaz score, have been shown to have excellent validity and reliability in the ENT patient population. These instruments can be used to document the initial dysphagia or dysphonia severity and monitor the treatment response in people with a wide array of swallowing and voice disorders.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing ACDF (single or multi-level) for the treatment of cervical radiculopathy or myelopathy
* All subjects must have given signed, informed consent prior to registration on study.

Exclusion Criteria:

* Patients undergoing revision surgery, any operations for trauma, infection, tumor
* Patients with general metabolic diseases such as rheumatoid arthritis, diabetes, chronic heart and renal diseases.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Medicine Department of Orthopaedic Surgery, Chicago, Illinois, United States

REFERENCES:
- [Background] Fountas KN, Kapsalaki EZ, Nikolakakos LG, Smisson HF, Johnston KW, Grigorian AA, Lee GP, Robinson JS Jr. Anterior cervical discectomy and fusion associated complications. Spine (Phila Pa 1976). 2007 Oct 1;32(21):2310-7. doi: 10.1097/BRS.0b013e318154c57e. PMID 17906571
- [Background] Sanfilippo JA Jr, Lim MR, Jacoby SM, Laterra R, Harrop JS, Vaccaro AR, Hilibrand AS, Anderson DG, Albert TJ. "Normal" prevertebral soft tissue swelling following elective anterior cervical decompression and fusion. J Spinal Disord Tech. 2006 Aug;19(6):399-401. doi: 10.1097/00024720-200608000-00004. PMID 16891973
- [Background] Pedram M, Castagnera L, Carat X, Macouillard G, Vital JM. Pharyngolaryngeal lesions in patients undergoing cervical spine surgery through the anterior approach: contribution of methylprednisolone. Eur Spine J. 2003 Feb;12(1):84-90. doi: 10.1007/s00586-002-0495-6. Epub 2002 Dec 4. PMID 12592551
- [Background] Lee SH, Kim KT, Suk KS, Park KJ, Oh KI. Effect of retropharyngeal steroid on prevertebral soft tissue swelling following anterior cervical discectomy and fusion: a prospective, randomized study. Spine (Phila Pa 1976). 2011 Dec 15;36(26):2286-92. doi: 10.1097/BRS.0b013e318237e5d0. PMID 22020609
- [Background] McAfee PC, Cappuccino A, Cunningham BW, Devine JG, Phillips FM, Regan JJ, Albert TJ, Ahrens JE. Lower incidence of dysphagia with cervical arthroplasty compared with ACDF in a prospective randomized clinical trial. J Spinal Disord Tech. 2010 Feb;23(1):1-8. doi: 10.1097/BSD.0b013e31819e2ab8. PMID 20051917
- [Background] Belafsky PC, Mouadeb DA, Rees CJ, Pryor JC, Postma GN, Allen J, Leonard RJ. Validity and reliability of the Eating Assessment Tool (EAT-10). Ann Otol Rhinol Laryngol. 2008 Dec;117(12):919-24. doi: 10.1177/000348940811701210. PMID 19140539

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | IV Steroid | Local Steroid
Started | 24 | 27 | 29
Completed | 21 | 25 | 29
Not Completed | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | IV Steroid | Local Steroid | Total
Number analyzed (Participants) | 21 | 25 | 29 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 20 | 23 | 58
  >=65 years | 6 | 5 | 6 | 17
Age, Continuous [Mean (Full Range); unit: years] | 54 [31 to 76] | 51.6 [28 to 81] | 55.6 [40 to 78] | 53.7 [28 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 14 | 35
  Male | 11 | 14 | 15 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0
  Unknown or Not Reported | 21 | 25 | 29 | 75
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 21 | 25 | 29 | 75
Region of Enrollment [Number; unit: participants]
  United States | 21 | 25 | 29 | 75

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Reporting Dysphagia/Severe Dysphagia Through EAT-10 From Baseline Through 1 Year Post-Op
Description: Outcome measure used to measure the incidence and severity of postoperative trouble swallowing. Summative score of 10 questions (range 0-40) with each question scored 0-4 with higher scores indicating greater severity/frequency of difficulty or disability reported by the patient for the indicated activity; EAT-10 >3 = dysphagia & EAT-10 >15 = severe dysphagia
Time Frame: baseline, post op day 1, post op 2 weeks, post op 6 weeks, post op 3 months, post op 6 months, and post op 1 year.
Population: All discrepancies between analyzed group participant totals and individual time point participant totals are due lack of patient response for follow-up data for the given time point despite multiple contact attempts by the research team
Measure: Number; unit: percentage
Arm/Group | Control Group | IV Steroid | Local Steroid
Number analyzed (Participants) | 21 | 25 | 29
percentage
  Baseline Dysphagia | 9.52 | 16.00 | 10.34
  Baseline Severe Dysphagia | 0 | 0 | 0
  1 Day Post Op Dysphagia: number analyzed (Participants) | 21 | 25 | 28
  1 Day Post Op Dysphagia | 76.19 | 68.00 | 61.90
  1 Day Post Op Severe Dysphagia: number analyzed (Participants) | 21 | 25 | 28
  1 Day Post Op Severe Dysphagia | 38.09 | 32.00 | 17.85
  2 wk. Post Op Dysphagia: number analyzed (Participants) | 20 | 25 | 29
  2 wk. Post Op Dysphagia | 50.00 | 48.00 | 27.58
  2 wk. Post Op Severe Dysphagia: number analyzed (Participants) | 20 | 25 | 29
  2 wk. Post Op Severe Dysphagia | 20.00 | 16.00 | 0.00
  6 wk. Post Op Dysphagia: number analyzed (Participants) | 21 | 23 | 29
  6 wk. Post Op Dysphagia | 38.09 | 34.78 | 17.24
  6 wk. Post Op Severe Dysphagia: number analyzed (Participants) | 21 | 23 | 29
  6 wk. Post Op Severe Dysphagia | 28.57 | 0.00 | 0.00
  3 mo. Post Op Dysphagia: number analyzed (Participants) | 20 | 23 | 29
  3 mo. Post Op Dysphagia | 20.00 | 8.69 | 6.89
  3 mo. Post Op Severe Dysphagia: number analyzed (Participants) | 20 | 23 | 29
  3 mo. Post Op Severe Dysphagia | 10.00 | 0.00 | 0.00
  6 mo. Post Op Dysphagia: number analyzed (Participants) | 19 | 24 | 29
  6 mo. Post Op Dysphagia | 21.05 | 8.33 | 13.79
  6 mo. Post Op Severe Dysphagia: number analyzed (Participants) | 19 | 24 | 29
  6 mo. Post Op Severe Dysphagia | 0.00 | 0.00 | 0.00
  1 yr. Post Op Dysphagia: number analyzed (Participants) | 19 | 23 | 29
  1 yr. Post Op Dysphagia | 21.05 | 0.00 | 6.89
  1 yr. Post Op Severe Dysphagia: number analyzed (Participants) | 19 | 23 | 29
  1 yr. Post Op Severe Dysphagia | 10.52 | 0.00 | 0.00

2. Primary Outcome: Percentage of Patients Reporting Abnormal Vocal Handicap Measured by the VHI-10 From Baseline Through 1 Year Post-Op
Description: Outcome measure used to measure the incidence and severity of postoperative trouble with hoarseness of voice; summative score of 10 questions (range 0-40) with each question scored 0-4 with higher scores indicating greater severity/frequency of disability or handicap reported by the patient. Reported as a percentage of patients in each group reporting an 'abnormal' VHI-10 score defined as a summative score >11
Time Frame: baseline, post op day 1, post op 2 weeks, post op 6 weeks, post op 3 months, post op 6 months, and post op 1 year.
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Control Group | IV Steroid | Local Steroid
Number analyzed (Participants) | 21 | 25 | 29
percentage of patients
  Baseline Abnormal VHI-10 | 9.52 | 8.00 | 3.44
  1 Day Post Op Abnormal VHI-10: number analyzed (Participants) | 21 | 25 | 28
  1 Day Post Op Abnormal VHI-10 | 4.76 | 4.00 | 3.57
  2 wk. Post Op Abnormal VHI-10: number analyzed (Participants) | 20 | 25 | 29
  2 wk. Post Op Abnormal VHI-10 | 10.00 | 20.00 | 0.00
  6 wk. Post Op Abnormal VHI-10: number analyzed (Participants) | 21 | 23 | 29
  6 wk. Post Op Abnormal VHI-10 | 9.52 | 8.69 | 3.44
  3 mo. Post Op Abnormal VHI-10: number analyzed (Participants) | 20 | 23 | 29
  3 mo. Post Op Abnormal VHI-10 | 10.00 | 4.34 | 0.00
  6 mo. Post Op Abnormal VHI-10: number analyzed (Participants) | 19 | 24 | 29
  6 mo. Post Op Abnormal VHI-10 | 10.53 | 8.33 | 3.44
  1 yr. Post Op Abnormal VHI-10: number analyzed (Participants) | 19 | 23 | 29
  1 yr. Post Op Abnormal VHI-10 | 10.53 | 8.33 | 0.00

3. Primary Outcome: Neck Disability Index (NDI) Mean Percentage Score From Baseline Through 1 Year Post Op
Description: Outcome measure used to measure for neck pain that includes personal care, lifting, reading, headaches, concentration, work, driving, sleeping and recreation. Summative scores for 10 questions (range 0-50) with each question scored 0-5 where higher scores for each question indicates greater extent of disability/difficulty for the associated activity. Reported as a mean percentage + standard deviation of difficulty/disability experienced by the patient.
Time Frame: Obtained at baseline, post op day 1, post op 2 weeks, post op 6 weeks, post op 3 months, post op 6 months, and post op 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of disability/difficulty
Arm/Group | Control Group | IV Steroid | Local Steroid
Number analyzed (Participants) | 21 | 25 | 29
percentage of disability/difficulty
  Baseline NDI | 40 (19) | 34 (18) | 35 (19)
  1 Day Post Op NDI: number analyzed (Participants) | 21 | 25 | 28
  1 Day Post Op NDI | 27 (14) | 28 (16) | 27 (18)
  2 wk. Post Op NDI: number analyzed (Participants) | 20 | 25 | 29
  2 wk. Post Op NDI | 31 (20) | 24 (15) | 20 (16)
  6 wk. Post Op NDI: number analyzed (Participants) | 21 | 23 | 29
  6 wk. Post Op NDI | 23 (19) | 21 (15) | 24 (19)
  3 mo. Post Op NDI: number analyzed (Participants) | 20 | 23 | 29
  3 mo. Post Op NDI | 14.6 (40) | 11.1 (23.3) | 10 (23.5)
  6 mo. Post Op NDI: number analyzed (Participants) | 19 | 24 | 29
  6 mo. Post Op NDI | 23 (19) | 21 (15) | 24 (19)
  1 yr. Post Op NDI: number analyzed (Participants) | 19 | 23 | 29
  1 yr. Post Op NDI | 22.2 (33.6) | 4.0 (18) | 6.0 (26)

4. Primary Outcome: Median Visual Analog Scale Pain Score for Patients From Baseline Through 1 Year Post Op
Description: Most commonly utilized pain scale; scored 0-10 with higher values indicating increased severity of pain experienced by the patient
Time Frame: Obtained at baseline, post op day 1, post op 2 weeks, post op 6 weeks, post op 3 months, post op 6 months, and post op 1 year; analyzed for all time points through 6 months post op
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Score on a scale
Arm/Group | Control Group | IV Steroid | Local Steroid
Number analyzed (Participants) | 21 | 25 | 29
Score on a scale
  VAS Pain Score (Baseline) | 8.0 [6.00 to 9.00] | 8.0 [6.00 to 9.00] | 7.0 [4.00 to 9.00]
  VAS Pain Score (1 Day Post Op): number analyzed (Participants) | 21 | 25 | 28
  VAS Pain Score (1 Day Post Op) | 7.00 [6.50 to 9.00] | 6.00 [3.00 to 9.00] | 6.00 [3.00 to 7.00]
  VAS Pain Score (2 wk. Post Op): number analyzed (Participants) | 20 | 25 | 29
  VAS Pain Score (2 wk. Post Op) | 6.00 [5.00 to 8.00] | 4.00 [3.00 to 6.00] | 4.00 [3.00 to 6.00]
  VAS Pain Score (6 wk. Post Op): number analyzed (Participants) | 21 | 23 | 29
  VAS Pain Score (6 wk. Post Op) | 5.00 [3.00 to 8.00] | 4.00 [2.00 to 5.50] | 5.00 [3.00 to 7.00]
  VAS Pain Score (3 mo. Post Op): number analyzed (Participants) | 20 | 23 | 29
  VAS Pain Score (3 mo. Post Op) | 4.5 [1.75 to 7.00] | 3.0 [1.00 to 4.00] | 3.00 [2.00 to 5.00]
  VAS Pain Score (6 mo. Post Op): number analyzed (Participants) | 19 | 24 | 29
  VAS Pain Score (6 mo. Post Op) | 5.0 [3.00 to 8.00] | 4.0 [2.00 to 5.50] | 5.00 [3.00 to 7.00]
  VAS Pain Score (1 yr. Post Op): number analyzed (Participants) | 19 | 23 | 29
  VAS Pain Score (1 yr. Post Op) | 4.0 [1.00 to 6.00] | 2.0 [1.00 to 4.00] | 1.0 [1.00 to 5.00]

5. Primary Outcome: Percentage of Patients Reporting Mild/Moderate/Severe Dysphagia From Baseline Through 1 Year Post Op Measured With Bazaz Dysphagia Score
Description: Outcome measure used to measure the incidence and severity of postoperative trouble swallowing
Time Frame: Evaluated at baseline, post op day 1, post op 2 weeks, post op 6 weeks, post op 3 months, post op 6 months, and post op 1 year
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Control Group | IV Steroid | Local Steroid
Number analyzed (Participants) | 21 | 25 | 29
percentage of patients
  Baseline Bazaz Score (Mild or Greater) | 4.76 | 0.00 | 6.89
  Baseline Bazaz Score (Moderate-Severe) | 0.00 | 0.00 | 0.00
  1 Day Post Op Bazaz Score (Mild or Greater): number analyzed (Participants) | 21 | 25 | 28
  1 Day Post Op Bazaz Score (Mild or Greater) | 61.90 | 44.00 | 50.00
  1 Day Post Op Bazaz Score (Moderate-Severe): number analyzed (Participants) | 21 | 25 | 28
  1 Day Post Op Bazaz Score (Moderate-Severe) | 33.33 | 24.00 | 7.14
  2 wk. Post Op Bazaz Score (Mild or Greater): number analyzed (Participants) | 20 | 25 | 29
  2 wk. Post Op Bazaz Score (Mild or Greater) | 30.00 | 16.00 | 13.79
  2 wk. Post Op Bazaz Score (Moderate-Severe): number analyzed (Participants) | 20 | 25 | 29
  2 wk. Post Op Bazaz Score (Moderate-Severe) | 15.00 | 16.00 | 0.00
  6 wk. Post Op Bazaz Score (Mild or Greater): number analyzed (Participants) | 21 | 23 | 29
  6 wk. Post Op Bazaz Score (Mild or Greater) | 28.57 | 17.39 | 6.89
  6 wk. Post Op Bazaz Score (Moderate-Severe): number analyzed (Participants) | 21 | 23 | 29
  6 wk. Post Op Bazaz Score (Moderate-Severe) | 23.80 | 8.69 | 0.00
  3 mo. Post Op Bazaz Score (Mild or Greater): number analyzed (Participants) | 20 | 23 | 29
  3 mo. Post Op Bazaz Score (Mild or Greater) | 15.00 | 13.04 | 13.79
  3 mo. Post Op Bazaz Score (Moderate-Severe): number analyzed (Participants) | 20 | 23 | 29
  3 mo. Post Op Bazaz Score (Moderate-Severe) | 15.00 | 0.00 | 0.00
  6 mo. Post Op Bazaz Score (Mild or Greater): number analyzed (Participants) | 19 | 24 | 29
  6 mo. Post Op Bazaz Score (Mild or Greater) | 15.78 | 8.33 | 13.79
  6 mo. Post Op Bazaz Score (Moderate-Severe): number analyzed (Participants) | 19 | 24 | 29
  6 mo. Post Op Bazaz Score (Moderate-Severe) | 5.26 | 0.00 | 0.00
  1 yr. Post Op Bazaz Score (Mild or Greater): number analyzed (Participants) | 19 | 23 | 29
  1 yr. Post Op Bazaz Score (Mild or Greater) | 15.78 | 0.00 | 3.44
  1 yr. Post Op Bazaz Score (Moderate-Severe): number analyzed (Participants) | 19 | 23 | 29
  1 yr. Post Op Bazaz Score (Moderate-Severe) | 5.26 | 0.00 | 3.44

ADVERSE EVENTS:
Time Frame: 1 year
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | Control Group | IV Steroid | Local Steroid
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/91/NCT02577991/Prot_SAP_000.pdf
  • Informed Consent Form (2015-12-21): https://cdn.clinicaltrials.gov/large-docs/91/NCT02577991/ICF_001.pdf